CLINICAL TRIAL: NCT01837342
Title: Multicenter Randomized Study Comparing Morbidity and Quality of Life Associated in the Treatment by Surgical Resection and the Conservative Treatment, After Favorable Evolution of Purulent Peritonitis That Originates From Diverticulitis Treated by Mini-invasive Surgery.
Brief Title: Multicenter Study Comparing Morbidity and Quality of Life Associated in the Treatment by Surgical Resection and the Conservative Treatment, After Favorable Evolution of Purulent Peritonitis That Originates From Diverticulitis Treated by Mini-invasive Surgery
Acronym: SIGMOIDITE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5061
Record Dates: First submitted 2012-11-26; First posted 2013-04-23 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Peritonitis; Diverticulitis
MeSH Terms: conditions — Peritonitis; Diverticulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sigmoidectomy arm (Other): Standard of care arm : sigmoid reserction after randomisation
  Interventions: Procedure: Surgical reserction
- Control arm (Experimental): laproscopic drainage and washing
  Interventions: Other: Radiological percutaneous drainage and washing drainage

INTERVENTIONS:
Procedure: Surgical reserction
  Arms: Sigmoidectomy arm
Other: Radiological percutaneous drainage and washing drainage
  Arms: Control arm

SUMMARY:
Sigmoid diverticular diseases is a pathologie frequent in patients above 60 years old. A person with diverticulosis may have few or no symptoms. When a diverticulum ruptures and infection sets in around the diverticulum the condition is called diverticulitis. An individual suffering from diverticulitis may have abdominal pain, abdominal tenderness, and fever. Bleeding originates from a diverticulum, it is called diverticular bleeding. Frequent hospitalisations as a result of the evolution of purulent peritonitis that originates from diverticulitis treated by mini-invasive surgery results.

Radiological percutaneous drainage and washing of the abdominal cavity during laparoscopic generalized purulent peritonitis of diverticular origin have been identified as therapeutic options by HAS (French health authorities), followed by second stage resection-anastomosis under elective surgery. It has been observed in patients that if only drainage and washing are performed (without resection), then the morbidity (10%) and mortality (1.5%) rates are much lower than usual rates (after resection) respectively 20-40% and 10-30%. Furthermore this reduces the risks of postoperatory complications.

Some studies have shown that the attitude of non-distance resection of the acute episode was associated with a recurrence rate of diverticulitis less than 5% recurrence without gravity. In addition, the morbidity associated with intervention sigmoid resection is around 30%.

The question arises in our daily practice, or not to propose systematic resection of sigmoid diverticulitis after an acute episode of severe purulent peritonitis or abscess types supported initially by minimally invasive.

The primary objective of the study is to determine, after clinical improvement linked to conservative treatment of perforated diverticulitis Hinchey peritonitis stage II and III, if a conservative approach reduces morbidity compared with a cold sigmoid resection attitude as currently recommended.

The secondary objective of the study is to determine if conservative treatment reduces mortality, length of hospital stay compared with cumulative sigmoid diverticular disease and improves quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had an episode of sigmoid diverticulitis as a result of pelvic or purulent peritonitis (Hinchey stage II and III) complications and treated by conservative treatment such as per cutaneous radiological drainage or laparoscopic-assisted per cutaneous drainage.
* Male and female individuals aged from 18 to 65 years old (both ages included).
* Absence of contra-indication for surgery ASA Score ≤3
* Participants must have signed informed consent document indicating that they understand the purpose and procedures required for the study and are willing to participate in the study and comply with the study procedures and restrictions
* Patients will sign an informed consent after haven been informed of the results of the previous medical visit.
* Patients must be affiliated with, or a beneficiary of a social security system

Exclusion Criteria:

* Subjects in the exclusion period (haven participated in a previous trial or an ongoing trial )
* Contra- indication to surgery
* ASA Score >3
* Past history of evolutive neoplasm,
* Subjects unable to consent (case of emergency, subjects having difficulties in understanding)
* Patients for which consultation visits will not be possible (e.g. tourists and people who cannot stay above 18 months in France).
* Pregnant and breastfeeding women
* Subjects under tutorship or curator ship
* Subjets under judicial protection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-11; Primary Completion 2017-08 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Determine which of the two aproaches: the conservative treatment or sigmoid resection reduces morbidity | 2 years
  The primary endpoint is the composite as predictable morbidity is different between groups. It is the occurrence of a disease episode in connection with diverticulosis or its treatment: recurrence of diverticulitis, the need for intervention in the sigmoid resection group drawn for a conservative attitude, postoperative complications Dindo stage ≥ II in case of sigmoid

SECONDARY OUTCOMES:
Determeine if the conservative treatment reduces mortaity and ameliorates quality of life diverticulitis patients | 2 years
  The secondary endpoints were mortality, the number and duration of cumulative report with sigmoid diverticular disease hospitalization, quality of life (SF-36 questionnaire, and QLQ CR29)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine ARVIEUX, MD,PHD, Principal Investigator — Clinique Universitaire de Chirurgie Digestive et de l'Urgence, CHU de Grenoble, BP 217; Cécile BRIGAND, MD, PHD, Study Chair — Chirurgie générale et digestive, Hôpital de Hautepierre, 67098 Strasbourg Cedex; Sébastien DAN, MD, Principal Investigator — Chirurgie Digestive, Centre Hospitalier Emile Muller,20, avenue de Dr R Laennec; David GUINIER, MD, Principal Investigator — Service de chirurgie digestive,Centre Hospitalier Bretagne Sud, 56100 Lorient; Mehdi KAROUI, MD, Principal Investigator — Chirurgie digestive et hépato-bibliaire, Hôpital Henri Mondor AP-HP,Créteil; Christophe MARIETTE, MD,PHD, Principal Investigator — chirurgie digestive et générale, Hôpital C Huriez ,Place de Verdun ,59037 Lille Cedex; MSIKA Simon, MD, Principal Investigator — Chirurgie digestive, Hôpital, Louis Mourier APHP, 178 rue des renouillers, 92700 Colombes; MUSCARI Fabrice, MD, PHD, Principal Investigator — Chirurgie Générale et Digestive, CHU RANGUEIL Avenue Jean, Poulhes 31054 - TOULOUSE CEDEX; Marc POCARD, MD, PHD, Principal Investigator — Unité clinique de chirurgie digestive, Hopital Lariboisière, 2 rue Ambroise Paré, 75475 Paris cedex 10; REGIMBEAU Jean Marc, MD, Principal Investigator — CHU Amiens Nord Place Victor, Pauchet 80054 Amiens; Didier RIO, MD, Principal Investigator — Service de chirurgie digestive et viscérale, Centre Hospitalier Bretagne Atlantique, 20 bd du général Guillaudot, 56000 Vannes; Karim SLIM, MD,PHD, Principal Investigator — Service de chirurgie digestive Hotel Dieu, Bd Léon Malfreyt; Bertrand SUC, MD, Principal Investigator — Chirurgie Générale et Digestive du Pr Fourtanier,Centre Hospitalier Universitaire de TOULOUSE - RANGUEIL Avenue Jean Poulhes 31054 - TOULOUSE CEDEX
Locations (14):
- France (14):
  - Chirurgie générale et digestive,Hôpital de Hautepierre,, Strasbourg, Alsace
  - Clinique Universitaire de Chirurgie Digestive et de l'Urgence, Grenoble, CHU de Grenoble
  - Chirurgie Digestive, Centre Hospitalier Emile Muller, 20, avenue de Dr R Laennec, Mulhouse, Mulhouse
  - Chirurgie générale et digestive,Hôpital de Hautepierre,, Hôpital de Hautepierre, Strasbourg Cedex
  - CHU Amiens Nord Place Victor Pauchet, Amiens
  - Service de chirurgie digestive Hotel Dieu, Clermont-Ferrand
  - Chirurgie digestive, Hôpital Louis Mourier APHP, 178 rue des renouillers, Colombes
  - chirurgie digestive et générale, Hôpital C Huriez Place de Verdun, Lille
  - Service de chirurgie digestiveCentre Hospitalier Bretagne Sud, Lorient
  - Unité clinique de chirurgie digestive, Hopital Lariboisière, 2 rue Ambroise Paré, Paris
  - Chirurgie digestive et hépato-bibliaire,Hôpital Pitié Salpêtrière, Paris
  - Chirurgie Générale et Digestive du Pr Fourtanier,Centre Hospitalier Universitaire, Toulouse
  - Chirurgie Générale et Digestive, CHU RANGUEIL Avenue Jean Poulhes 31054, Toulouse
  - Centre Hospitalier Bretagne Atlantique, 20 bd du général Guillaudot,, Vannes